CLINICAL TRIAL: NCT02615782
Title: A Randomized, Open-label, Oral Single Dosing, Two-way Crossover Clinical Trial to Evaluate the Effects of Food on the Bioavailability of CKD-397 After a Single Oral Dose in Healthy Male Subjects
Brief Title: A Clinical Trial to Evaluate the Effects of Food on the Bioavailability of CKD-397 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 150FDI15031
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Benign Prostatic Hypertrophy (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A group (Experimental): 1. Period 1: CKD-397 1T single oral administration under fasting condition
  2. Period 2: CKD-397 1T single oral administration under fed condition (high fat meals)
  Interventions: Drug: CKD-397
- B group (Experimental): 1. Period 1: CKD-397 1T single oral administration under fed condition (high fat meals)
  2. Period 2: CKD-397 1T single oral administration under fasting condition
  Interventions: Drug: CKD-397

INTERVENTIONS:
Drug: CKD-397 — CKD-397 1T single oral administration under fasting condition or fed condition(high fat meals)
  Other Names: Tamsulosin HCl/Tadalafil 0.2/5mg; HARNAL-D Tab. 0.2mg + Cendom® Tab. 5mg

SUMMARY:
This study is a randomized, open-label, oral single dosing, two-way crossover clinical trial to evaluate the effects of food on the bioavailability of CKD-397 after a single oral dose in healthy male subjects

DETAILED DESCRIPTION:
To healthy male subjects of sixteen(16), following treatments are administered dosing in each period and wash-out period is a minimum of 10 days.

Treatment A: CKD-397 1T under Fasting condition Treatment B: CKD-397 1T under Fed condition (high fat meals). Pharmacokinetic blood samples are collected up to 72hrs. Safety and pharmacokinetic are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject older than 19 years at the time of screening.
2. Subjects who BMI more than 17.5kg/m2 and less than 30.5kg/m2 and weight more than 55kg
3. Subjects who signed the informed consent form after understanding fully to hear a detailed explanation in the clinical trial

Exclusion Criteria:

1. Subjects who have a history of blood, kidneys, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurological or allergic diseases that is clinically significant (Except untreated asymptomatic seasonal allergies at the time of administration)
2. Subjects who have a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption.
3. Subjects who show AST or AST > 2 times upper limit of normal range or eGFR < 60 mL/min/1.73m2
4. Subjects who drink Alcohol > 210g/week within 6 months prior to the screening.
5. Subjects who take the medication involved in other clinical trials or bioequivalence tests within three months before the first dose medication characters.
6. Subjects who show Systolic Blood Pressure ≤100 or ≥150 mmHg or Diastolic Blood Pressure ≤60 or ≥100 mmHg at screening
7. Subjects who have orthostatic hypotension
8. Subjects who have history of drug abuse or drug abuse positive at screening
9. Subjects who treated with metabolizing enzyme inducers or inhibitors such as barbitals within 30days prior to the first dosing.
10. Smoker ( ≥ 20cigarettes/day)
11. Subjects who takes ETC or herb medicine within two weeks or OTC or vitamin supplement within 1 week before the first IP administration
12. Subjects who do the whole blood donation within two months or component blood donation within 1month prior to the first dosing or receive blood transfusion within 1month prior to the first dosing
13. Subjects who can increase risk due to clinical test and administration of drugs or has Severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of test results
14. Subjects who take organic nitrate medicine regularly or intermittently
15. Patients with genetic degenerative retinal disease including retinitis pigmentosa
16. Subjects who have hypersensitivity to medicines including tadalafil/tamsulosin component or any other medicines(aspirin, antibiotics etc.) or medical history of clinically significant hypersensitivity
17. Patients who lost sight of one eye by Non-arteritic anterior ischemic optic neuropathy(NAION)
18. Subjects with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
19. Subjects who use a trustworthy method of contraception
20. Subjects who is not able to comply with guidelines described in the protocol
21. Subjects who is determined by investigator's decision including laboratory test result or another reason as unsuitable for clinical trial participation

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUClast of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs
Cmax of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs

SECONDARY OUTCOMES:
AUCinf of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs
Tmax of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs
t1/2 of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs
CL/F of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs
Vd/F of Tadalafil and Tamsulosin | 0(Pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 and 72hrs

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyu Park, MD, PhD, Principal Investigator — Domg-A University Hospital
Locations (1):
- Dong-A University Hospital, Seo-gu, Busan, South Korea